CLINICAL TRIAL: NCT00368173
Title: IGF-I/IGFBP-3 Therapy in Children and Adolescents With Growth Hormone Insenitivity Syndrome (GHIS) Such as Laron Syndrome
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Insmed Incorporated (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INSM-110-303
Record Dates: First submitted 2006-08-23; First posted 2006-08-24 (Estimated); Last update posted 2012-09-13 (Estimated); Status verified 2012-09

CONDITIONS: Growth Hormone Insensitivity Syndrome (GHIS); Laron Syndrome
MeSH Terms: conditions — Laron Syndrome | interventions — Insulin-Like Growth Factor I

INTERVENTIONS:
Drug: rhIGF-I/rhIGFBP-3

SUMMARY:
STUDY OBJECTIVE

To evaluate the safety, tolerability, and efficacy, as growth velocity (statural growth), of rhIGF-I/rhIGFBP-3 administered for 12 months in pre-pubertal children and adolescents with GHIS.

STUDY DESIGN

This study is an open-label, multi-center clinical trial to evaluate the safety and effectiveness of rhIGF-I/rhIGFBP-3 to increase rate of growth when administered once daily for 12 months in children and adolescents with growth hormone insensitivity syndrome (GHIS) such as Laron Syndrome. At the end of the initial twelve-month treatment period, additional safety and long-term efficacy data will be assessed in a second 12 month treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of GHIS such as Laron syndrome,
2. 2 - 18 years of age,
3. Height less than or equal to -3SD for age,
4. Pre-pubertal, defined as Tanner breast stage 1 or testis volume <4mL

Exclusion Criteria:

1. Children in puberty,
2. Diagnosed malignancy,
3. A diagnosis of diabetes mellitus

Ages: 2 Years to 18 Years | Sex: All
Age Groups: Child, Adult

CONTACTS AND LOCATIONS:
Locations (15):
- Robert Rapaport, MD, New York, New York, United States
- Argentina (2):
  - Dr. Alicia Belgorosky, Buenos Aires
  - Dr. Christina Bazan, San Miguel de Tucumán
- Dr. Bruce King, Newcastle, Australia
- Dr. Durval Damiani, São Paulo, Brazil
- Dr. Kwok-leung NG, Hong Kong, China
- Dr. Mohamed EL Kholy, Cairo, Egypt
- Professor Annette Greuters, Berlin, Germany
- Tiosano Dov, Haifa, Israel
- Maria Carolina Salerno, Naples, Italy
- Dr. Hilde Bjorndalen, Oslo, Norway
- Dr. Carlos del Aguila, Lima, Peru
- Dr. Magdalena Paskova, Košice, Slovakia
- Professor Nursen Yordam, Ankara, Turkey (Türkiye)
- Dr. Cecilia Camacho-Hubner, London, United Kingdom